CLINICAL TRIAL: NCT06063174
Title: Identifying Social, Molecular, & Immunological Processes for Mitigating Toxic Stress & Enhancing Personalized Resilience
Brief Title: Stress & Resilience Study
Acronym: CALSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Stanford University (Other); University of California, San Francisco (Other); California Initiative to Advance Precision Medicine (Other)
Responsible Party: Principal Investigator, George M. Slavich, PhD, Lead Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPR21101
Record Dates: First submitted 2023-09-06; First posted 2023-10-02 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-09

CONDITIONS: Stress; Stress, Psychological; Stress, Physiological; Stress, Emotional; Stress Reaction
Keywords: Stress; Immunology; Psychosocial; Clinical; Resilience
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (4):
- Baseline-Only (No Intervention): Baseline-only condition will be cross-sectional, and participants will be only completing the first portion of the study. Participants in this arm will be asked to wear a research-grade smartwatch for at least one week and complete the baseline package at one time point which includes self-reported questionnaires, micro-blood collection, and optional stool collection.
- Active Control (Active Comparator): Active control condition will be longitudinal. Participants in this arm will be asked to wear a research-grade smartwatch for at least 24 weeks and complete the baseline package as well as two follow-ups over a period of 24 weeks. After completing the baseline package, participants in the active control group will receive a 12 week psychoeducation training on stress and health called the Environmental Education Program.
  Interventions: Behavioral: Education Program
- Nonactive Control (No Intervention): Nonactive control condition will be longitudinal. Participants in this arm will be asked to wear a research-grade smartwatch for at least 24 weeks and complete the baseline package as well as two follow-ups over a period of 24 weeks. After completing the baseline package, participants in the nonactive control group will not be receiving any forms of intervention. Participants in this program called the Follow-up Program will be tracked over 12 weeks in parallel to participants receiving an intervention and another 12 weeks after.
- CAL STAR Personalized Intervention (Experimental): CAL STAR Personalized Intervention condition will be longitudinal. Participants in this arm will be asked to wear a research-grade smartwatch for at least 24 weeks and complete the baseline package as well as two follow-ups over a period of 24 weeks. After completing the baseline package, participants will be assigned to one of the five CAL STAR Personalized Intervention training programs (Think Well, Be Well, Eat Well, Sleep Well, Move Well programs) depending on their score on a self-reported survey called Consequences of Stress Scale (CSS). Based on the CSS score, a participant will be assigned to one of the five programs to work on a domain that is dysregulated when they are stressed. When eligible for multiple, their availability to attend coaching sessions and preferences will be accounted for, or they will be randomly assigned to conditions for which they are eligible.
  Interventions: Behavioral: Think Well Program; Behavioral: Be Well Program; Behavioral: Eat Well Program; Behavioral: Sleep Well Program; Behavioral: Move Well Program

INTERVENTIONS:
Behavioral: Education Program — 12-week online psychoeducation program on environmental pollution exposures, the health impacts and sources of these exposures, and practical ways to reduce these exposures. Participants in the active control group will receive this form of intervention.
  Arms: Active Control
Behavioral: Think Well Program — 12-week online program in which participants learn to identify negative emotion and thinking patterns and participate in live online group coaching. Participants whose thinking style domain is dysregulated will be assigned to this intervention program.
  Arms: CAL STAR Personalized Intervention
Behavioral: Be Well Program — 12-week online program in which participants learn about the importance of social relationships, connectedness, and interpersonal conflicts, and participate in live online group coaching. Participants whose social relationship/conflict domain is dysregulated will be assigned to this intervention program.
  Arms: CAL STAR Personalized Intervention
Behavioral: Eat Well Program — 12-week online program in which participants learn about mindful eating and participate in live online group coaching. Participants whose diet domain is dysregulated will be assigned to this intervention program.
  Arms: CAL STAR Personalized Intervention
Behavioral: Sleep Well Program — 12-week online program in which participants learn about the importance of good sleep and participate in live online group coaching. Participants whose sleep domain is dysregulated will be assigned to this intervention program.
  Arms: CAL STAR Personalized Intervention
Behavioral: Move Well Program — 12-week online program in which participants learn about the importance of adequate physical activity for health and participate in live online group coaching. Participants whose physical activity domain is dysregulated will be assigned to this intervention program.
  Arms: CAL STAR Personalized Intervention

SUMMARY:
Goal 1: The investigators will quantify lifetime stress burden and examine mechanisms linking Adverse Childhood Experiences (ACEs) and health. The investigators will quantify the early life and total lifetime stress burden of a representative sample of about 725 adults (aged 18+) across northern and southern California. In addition, the investigators will examine how prior life stress exposure and current stress levels are associated with differences in psychosocial, immune, metabolic, physiologic, and clinical outcomes for all participants at baseline.

Goal 2: The investigators will develop and test a biopsychosocial intervention using existing programs, platforms, resources, and core components from trauma and resilience research that will target five stress-related domains (i.e., cognitive response style, social relationships, eating, sleep, and physical activity) using cognitive restructuring and mindfulness, interpersonal skills training, mindful eating training, sleep training, and behavioral activation/mobility training. The investigators will then assess the efficacy and acceptability of the intervention in about 425 high stress exposure participants from Goal 1. Following their baseline assessment, about 425 participants will be randomly assigned to receive for 12 weeks (a) personalized intervention, (b) environmental education (active control) or (c) nothing (non-active control). The investigators will also assess the efficacy of the personalized intervention by comparing changes in outcomes by condition from baseline (prior to randomization) to immediately after the intervention, and then again after 12 weeks following intervention completion. The interventions will be entirely online/remote.

DETAILED DESCRIPTION:
Aim 1: The investigators will quantify lifetime stress burden and examine mechanisms linking Adverse Childhood Experiences (ACEs) and health. The investigators will quantify the early life and total lifetime stress burden of a representative sample of about 725 adults (aged 18+) across California. In addition, the investigators will examine how prior life stress exposure and current stress levels are associated with differences in psychosocial, immune, metabolic, physiologic, and clinical outcomes for all participants at baseline.

Objective 1.1. Characterize associations between stress levels and psychosocial and clinical functioning by collecting self-report data from participants (see below) and by using any available electronic health records.

Objective 1.2. Examine cross-sectional relations between stress levels and physiological, biological, and behavioral processes using (1) immune and metabolic functioning assessed by non-invasive blood microsampling and the investigators' unique multi-omics approach, and (2) continuously monitored physiologic and behavioral functioning using smartwatches that have the ability to assess a variety of physiologic & behavioral processes (e.g., cardiac function, sleep, activity levels).

Objective 1.3. Develop a Personal Health Dashboard for processing data with an algorithm that will generate personalized results to inform individualized health risk assessments and provide an opportunity to deliver tailored clinical feedback and biopsychosocial resiliency training by targeting five key stress-related risk factors (see Aim 2).

Aim 2: Reduce ACEs-related health disparities by developing and testing a behavioral intervention for about 425 of the higher stress participants from Aim 1. To reduce negative stress-related effects and bolster resilience, the investigators will examine the acceptability and effectiveness of a 12 week, online, precision behavioral intervention.

Objective 2.1. Develop a behavioral intervention using existing programs, platforms, resources, and core components from trauma and resilience research that will target five stress-related domains (i.e., perceived stress, social relationships, diet, sleep, and physical activity) using cognitive restructuring and mindfulness, interpersonal skills training, personalized diet training, sleep training, and behavioral activation.

Objective 2.2. Assess the efficacy of the above-described intervention in about 425 high stress exposure participants from Goal 1. Following their baseline assessment, participants will be randomly assigned to receive (a) the personalized intervention (about 55 participants per stress-related domain), (b) stress & health psychoeducation/active control group, or (c) nonactive control group. For participants receiving the intervention, the investigators will identify each person's most dysregulated biobehavioral process using the comprehensive biopsychosocial data obtained from Goal 1, focusing on five major stress-related domains: cognitive response style, social relationships, eating, sleep, and physical activity. The investigators will pilot the use of online coach-assisted personalized interventions to target a dysregulated domain for each participant. The investigators will also assess the efficacy of the intervention by comparing changes in outcomes by condition from baseline (prior to randomization) to immediately after the intervention, and then again several months following intervention completion. The primary outcome of interest will be perceived stress (PSS-10). The secondary outcomes of the RCT include five domain specific surveys: the Five-Factor Mindfulness Scale short form (cognitive response style), Conflict Scale and UCLA Loneliness Scale (social relationship domain), Salzburg Stress Eating Scale (eating domain), Insomnia Severity Index (sleeping domain), and International Physical Activity Questionnaire short form (IPAQ, physical activity domain). Exploratory outcomes include the multiomics measures (including untargeted metabolomics, lipidomics, immune proteins, cytokines and the microbiome), physiological measures from the wearable device (i.e., heart rate variability), and continuous glucose monitoring measures.

ELIGIBILITY:
Inclusion Criteria:

* A participant must meet all of the following criteria to be eligible to participate in this study:

  1. Be able to understand and agree to comply with planned study procedures in English.
  2. Participants must be aged 18 or over.
  3. Participants must reside in the state of California.

Exclusion Criteria:

* A participant who meets any of the following criteria will be excluded from participation in this study:

History of disease(s):

1. Has a positive test result for human immunodeficiency virus (HIV) types 1 or 2 antibodies.
2. Has had a heart attack or stroke within the past year.
3. Has had and/or been treated for any type of cancer in the past two years.

Medication(s):

Participants who check off any of the following medications and/or treatment listed below over the past month will be excluded in the study.

1. Prednisolone (e.g., Omnipred, Pred Mild, Pred Forte, Orapred ODT, Veripred 20, Millipred DP)
2. Prednisone (e.g., Prednisone Intensol, Deltasone, Rayos)
3. Betamethasone (e.g., Celestone Soluspan, Sernivo, Diprolene AF, ReadySharp Betamethasone, Betaloan SUIK, Beta-1)
4. Dexamethasone (e.g., Ozurdex, Maxidex, DexPak 6 Day/10 day/13 Day, LoCort, ZonaCort, ReadySharp dexamethasone, DoubleDex)
5. Hydrocortisone (e.g., Hydrocort, Alphosyl, Aquacort, Cortef, Cortenema, and Solu-Cortef)
6. Methylprednisolone (e.g., Depo-Medrol, Solu-Medrol, Medrol, ReadySharp Methylprednisolone, P-Care D80, and P-Care D40)
7. Deflazacort (e.g., Emflaza)
8. Immunomodulators

   * Cyclosporine (Sandimmune, Neoral, Gengraf, Restasis MultiDose)
   * Tacrolimus (Protopic, Envarsus XR, Astagraf XL, Prograf)
   * Methotrexate (Rheumatrex, Trexall, Otrexup (PF), Xatmep, Rasuvo, Mexate, MTX)
   * Azathioprine (Immuran, Azasan)
   * Mercaptopurine (6-MP, Purinethol, Purixan)
   * Other Immunomodulators not listed above
9. Monoclonal antibody therapy

   * Infliximab (Remicade)
   * Etanercept (Enbrel, Benepali, Erelzi)
   * Adalimumab (Humira)
   * Secukinumab (Cosentyx)
   * Tofacitinib (Xeljanz)
   * Rituximab (Rituxan)
   * Other Monoclonal antibody therapy not listed above
10. Intravenous immunoglobulin treatment (IVIG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in PSS-10 | PSS-10 will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The primary endpoint will be the change in Perceived Stress Scale (PSS-10) score between the nonactive control, active control, and the treatment groups (combined) from screening to Follow-up 1 & 2. A meaningful clinically significant score in the PSS-10 score is a difference of 5 points. The range of the PSS-10 is 0-40, with higher scores indicating more perceived stress. As such PSS-10 change scores could range from -40 to 40. A positive PSS-10 change score indicates increased stress and is a negative outcome. A negative PSS-10 change score indicates decreased stress and is a positive outcome.

SECONDARY OUTCOMES:
Change in CSS subscale Score | Consequences of Stress scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific intervention risk score between screening and Follow-up 1 & 2 from the Consequences of Stress scale (CSS) within intervention groups. Each CSS subscale has a range of 3-21, with higher scores indicating more dysfunction. As such, CSS subscale change scores could be from -18 to 18. A positive CSS subscale change score indicates increased dysfunction and is a negative outcome. A negative CSS subscale change score indicates decreased dysfunction and is a positive outcome.
Change in Five-Factor Mindfulness Scale short form (cognitive response style domain) | Five-Factor Mindfulness scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific domain score between screening and Follow-up 1 & 2 from the Five Factor Mindfulness Scale (FFMS) partial short form within the cognitive response style group. The FFMS-15 short form was reduced to a 6-item questionnaire to include only non-judgement and non-reactivity subscales. The scale has a range of 6-30, which higher scores indicating increased mindfulness. FFMS change scores could be from -24 to 24. A positive FFMS scale change score indicates decreased mindfulness and is a negative outcome. A negative FFMS scale change score indicated increased mindfulness and is a positive outcome.
Change in Conflict Scale and UCLA Loneliness Scale (social relationship domain) | Five-Factor Mindfulness scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific domain score between screening and Follow-up 1 & 2 from the Conflict Scale and UCLA Loneliness Scale short form within the social relationship group. The revised Conflict Scale has a range of 6-42, with higher scores indicating more conflict. Conflict scale change scores could be from -36 to 36. A positive Conflict scale change score indicates increased conflict and is a negative outcome. A negative Conflict scale change score indicates decreased conflict and is a positive outcome. The UCLA Loneliness Scale has a range of 3-9, which higher score indicating more loneliness. UCLA Loneliness Scale change scores could be from -6 to 6. A positive UCLA Loneliness scale change score indicates increased loneliness and is a negative outcome. A negative UCLA Loneliness scale change score indicates decreased loneliness and is a positive outcome.
Change in Salzburg Stress Eating Scale (eating domain) | Salzburg Stress Eating scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific domain score between screening and Follow-up 1 & 2 from the Salzburg Stress Eating Scale (SSES) within the eating group. The scale has a range of 10-50, which higher scores indicating tendency to eat more when stressed, medium score indicating tendency to eat just as much as usual when stressed, and lower score indicating tendency to eat less when stressed. SSES change scores could be from -40 to 40. A mean score towards a medium mean score (=3) indicates tendency to eat just as much has usual when stressed and is a positive outcome. Higher or lower means indicate tendency to over and/or under eat and is a negative outcome.
Change in Insomnia Severity Index (sleeping domain) | Insomnia Severity Index scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific domain score between screening and Follow-up 1 & 2 from the Insomnia Severity Index (ISI) within the sleep group. The scale has a range of 0-28, which higher scores indicating increased insomnia or sleep issues. ISI scale change scores could be from -28 to 28. A positive ISI scale change score indicates increased insomnia and is a negative outcome. A negative FFMS scale change score indicated decreased insomnia and is a positive outcome.
Change in International Physical Activity Questionnaire short form (physical activity domain) | International Physical Activity Questionnaire scale will be assessed at all three time points during the baseline period (first 1-3 weeks of the study), follow-up1 (after 12-week intervention), and follow-up2 (at 24 week mark from baseline).
  The change in participants' specific domain score between screening and Follow-up 1 & 2 from the International Physical Activity Questionnaire (IPAQ) short form within the physical activity group. The scale has two forms of output from scoring. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). The continuous variable will be used for analysis purposes by estimating total MET minutes/week (range 0- 10080). MET minutes represent the amount of energy expended carrying out physical activity. Higher scores indicate increased level of physical activity and is a positive outcome. Lower scores indicate decreased levels of physical activity and is a negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: George M Slavich, PhD, Principal Investigator — University of California, Los Angeles; Michael P Snyder, PhD, Principal Investigator — Stanford University; Alicia F Lieberman, PhD, Principal Investigator — University of California, San Francisco; Shannon Thyne, MD, Principal Investigator — Los Angeles County Department of Public Health; Patricia E Lester, MD, Principal Investigator — University of California, Los Angeles; Atul J Butte, MD,PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Hughes K, Bellis MA, Hardcastle KA, Sethi D, Butchart A, Mikton C, Jones L, Dunne MP. The effect of multiple adverse childhood experiences on health: a systematic review and meta-analysis. Lancet Public Health. 2017 Aug;2(8):e356-e366. doi: 10.1016/S2468-2667(17)30118-4. Epub 2017 Jul 31. PMID 29253477
- [Background] California Department of Public Health and Department of Social Services. Adverse Childhood Experiences Data Report: Behavioral Risk Factor Surveillance System (BRFSS), 2011-2017: An Overview of Adverse Childhood Experiences in California. (2020). doi:10.48019/PEAM8812.
- [Background] Hargreaves MK, Mouton CP, Liu J, Zhou YE, Blot WJ. Adverse Childhood Experiences and Health Care Utilization in a Low-Income Population. J Health Care Poor Underserved. 2019;30(2):749-767. doi: 10.1353/hpu.2019.0054. PMID 31130549
- [Background] Birn RM, Roeber BJ, Pollak SD. Early childhood stress exposure, reward pathways, and adult decision making. Proc Natl Acad Sci U S A. 2017 Dec 19;114(51):13549-13554. doi: 10.1073/pnas.1708791114. Epub 2017 Dec 4. PMID 29203671
- [Background] Slavich GM. Social Safety Theory: A Biologically Based Evolutionary Perspective on Life Stress, Health, and Behavior. Annu Rev Clin Psychol. 2020 May 7;16:265-295. doi: 10.1146/annurev-clinpsy-032816-045159. Epub 2020 Mar 6. PMID 32141764
- [Background] Slavich GM, Way BM, Eisenberger NI, Taylor SE. Neural sensitivity to social rejection is associated with inflammatory responses to social stress. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14817-22. doi: 10.1073/pnas.1009164107. Epub 2010 Aug 2. PMID 20679216
- [Background] Cohodes EM, Kitt ER, Baskin-Sommers A, Gee DG. Influences of early-life stress on frontolimbic circuitry: Harnessing a dimensional approach to elucidate the effects of heterogeneity in stress exposure. Dev Psychobiol. 2021 Mar;63(2):153-172. doi: 10.1002/dev.21969. Epub 2020 Mar 29. PMID 32227350
- [Background] Gee DG, Casey BJ. The Impact of Developmental Timing for Stress and Recovery. Neurobiol Stress. 2015 Jan 1;1:184-194. doi: 10.1016/j.ynstr.2015.02.001. PMID 25798454
- [Background] Miller TR, Waehrer GM, Oh DL, Purewal Boparai S, Ohlsson Walker S, Silverio Marques S, Burke Harris N. Adult health burden and costs in California during 2013 associated with prior adverse childhood experiences. PLoS One. 2020 Jan 28;15(1):e0228019. doi: 10.1371/journal.pone.0228019. eCollection 2020. PMID 31990957
- [Background] Waehrer GM, Miller TR, Silverio Marques SC, Oh DL, Burke Harris N. Disease burden of adverse childhood experiences across 14 states. PLoS One. 2020 Jan 28;15(1):e0226134. doi: 10.1371/journal.pone.0226134. eCollection 2020. PMID 31990910
- [Background] Bhushan D, Kotz K, McCall J, etal. Road map for Resilience: The California Surgeon General's Report on Adverse Childhood Experiences, Toxic Stress, and Health.(2020). doi:10.48019/PEAM8812
- [Background] Giano Z, Wheeler DL, Hubach RD. The frequencies and disparities of adverse childhood experiences in the U.S. BMC Public Health. 2020 Sep 10;20(1):1327. doi: 10.1186/s12889-020-09411-z. PMID 32907569
- [Background] Dwyer-Lindgren L, Bertozzi-Villa A, Stubbs RW, Morozoff C, Mackenbach JP, van Lenthe FJ, Mokdad AH, Murray CJL. Inequalities in Life Expectancy Among US Counties, 1980 to 2014: Temporal Trends and Key Drivers. JAMA Intern Med. 2017 Jul 1;177(7):1003-1011. doi: 10.1001/jamainternmed.2017.0918. PMID 28492829
- [Background] Stork BR, Akselberg NJ, Qin Y, Miller DC. Adverse Childhood Experiences (ACEs) and Community Physicians: What We've Learned. Perm J. 2020;24:19.099. doi: 10.7812/TPP/19.099. Epub 2020 Jan 24. PMID 32069204
- [Background] Valderhaug TG, Slavich GM. Assessing Life Stress: A Critical Priority in Obesity Research and Treatment. Obesity (Silver Spring). 2020 Sep;28(9):1571-1573. doi: 10.1002/oby.22911. Epub 2020 Jul 29. PMID 32729167
- [Background] Chambers DA, Norton WE. The Adaptome: Advancing the Science of Intervention Adaptation. Am J Prev Med. 2016 Oct;51(4 Suppl 2):S124-31. doi: 10.1016/j.amepre.2016.05.011. Epub 2016 Jun 28. PMID 27371105
- [Background] Wang YA, Rhemtulla M. Power analysis for parameter estimates in structural equation modeling:A discussion and tutorial. Adv Methods Pract Psychol Sci. doi:10.31234/osf.io/pj67b
- [Background] Shields GS, Spahr CM, Slavich GM. Psychosocial Interventions and Immune System Function: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Psychiatry. 2020 Oct 1;77(10):1031-1043. doi: 10.1001/jamapsychiatry.2020.0431. PMID 32492090
- [Background] Kivimaki M, Steptoe A. Effects of stress on the development and progression of cardiovascular disease. Nat Rev Cardiol. 2018 Apr;15(4):215-229. doi: 10.1038/nrcardio.2017.189. Epub 2017 Dec 7. PMID 29213140
- [Background] Truelsen T, Nielsen N, Boysen G, Gronbaek M; Copenhagen City Heart Study. Self-reported stress and risk of stroke: the Copenhagen City Heart Study. Stroke. 2003 Apr;34(4):856-62. doi: 10.1161/01.STR.0000062345.80774.40. Epub 2003 Mar 13. PMID 12637696
- [Background] Slavich GM, Irwin MR. From stress to inflammation and major depressive disorder: a social signal transduction theory of depression. Psychol Bull. 2014 May;140(3):774-815. doi: 10.1037/a0035302. Epub 2014 Jan 13. PMID 24417575
- [Background] Chiang JJ, Park H, Almeida DM, Bower JE, Cole SW, Irwin MR, McCreath H, Seeman TE, Fuligni AJ. Psychosocial stress and C-reactive protein from mid-adolescence to young adulthood. Health Psychol. 2019 Mar;38(3):259-267. doi: 10.1037/hea0000701. PMID 30762405
- [Background] Weyh C, Kruger K, Strasser B. Physical Activity and Diet Shape the Immune System during Aging. Nutrients. 2020 Feb 28;12(3):622. doi: 10.3390/nu12030622. PMID 32121049
- [Background] Barton W, Penney NC, Cronin O, Garcia-Perez I, Molloy MG, Holmes E, Shanahan F, Cotter PD, O'Sullivan O. The microbiome of professional athletes differs from that of more sedentary subjects in composition and particularly at the functional metabolic level. Gut. 2018 Apr;67(4):625-633. doi: 10.1136/gutjnl-2016-313627. Epub 2017 Mar 30. PMID 28360096
- [Background] Adamantidis A, de Lecea L. Sleep and metabolism: shared circuits, new connections. Trends Endocrinol Metab. 2008 Dec;19(10):362-70. doi: 10.1016/j.tem.2008.08.007. Epub 2008 Oct 18. PMID 18938086